CLINICAL TRIAL: NCT04163237
Title: Study on Combined Immunotherapy and Targeted Therapy for Advanced Liver Cancer
Brief Title: Combined Immunotherapy and Targeted Therapy for Advanced Liver Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, TaoBai, Researcher, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GuangXiMU-HCC-PD1(2)
Record Dates: First submitted 2019-11-06; First posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Advanced Liver Cancer
MeSH Terms: interventions — Sorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-1 & Sorafenib (Experimental)
  Interventions: Drug: PD-1; Drug: Sorafenib
- Sorafenib (Other)
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: PD-1 — PD-1 (programmed death receptor 1), an important immunosuppressive molecule, is an immunoglobulin superfamily and is a membrane protein of 268 amino acid residues. It was originally cloned from apoptotic mouse T cell hybridoma 2B4.11. Immunomodulation targeting PD-1 has important implications for anti-tumor, anti-infective, anti- autoimmune diseases and organ transplant survival. Its ligand PD-L1 can also be used as a target, and the corresponding antibodies can also play the same role. PD-1 and PD-L1 bind to initiate programmed cell death of T cells, allowing tumor cells to gain immune escape.
  Arms: PD-1 & Sorafenib
Drug: Sorafenib — Sorafenib tosylate is a novel multi- target anti-tumor drug developed by Bayer Pharmaceuticals, Germany, which acts on both tumor cells and tumor blood vessels. It has a dual anti-tumor effect: it directly inhibits tumor cell proliferation by blocking RAF/MEK/ERK-mediated cell signaling pathways, and also by inhibiting VEGFR and platelet- derived growth factor (PDGF) receptors. Blocking the formation of tumor neovascularization, indirectly inhibiting the growth of tumor cells.

SUMMARY:
Liver cancer is a common malignant tumor in China, and its incidence rate ranks third and remains high. The treatment of liver cancer has made some progress in recent years, mainly the progress of radical treatment such as surgery and ablation. For liver cancer, due to the emergence of molecularly targeted drugs such as sorafenib and immunological checkpoint inhibitors, the systemic therapeutic effect of advanced liver cancer is improved, and the curative effect is further improved. In recent years, immunotherapy has become one of the clinical treatment options for cancer. T lymphocytes are a cell with cell killing ability in the immune system, and programmed death factor 1 (PD-1) is an important inhibitory receptor on the surface of T lymphocytes. It is known that the ligands of PD-1 are PD-L1 and PD-L2, and studies have found that a variety of tumor cells have high expression of PD-L1 ligand on the surface. At present, clinical research on target drugs for PD-1 has included dozens of solid tumors or hematological tumors. The results of clinical studies that have been completed and the interim results of some studies indicate that anti- PD-1 antibody drugs are more effective and safer than previous treatments. Patients with hepatocellular carcinoma (HCC) often undergo liver cancer resection, but the recurrence rate can reach 70% to 100%, which seriously affects the treatment outcome and long-term survival rate. Early recurrence of liver cancer is mainly related to the invasiveness of the tumor. Microvascular invasion, non-anatomical hepatectomy, AFP greater than 32 ng/ml, tumor diameter greater than 5 cm, and incomplete tumor capsule are risk factors for recurrence within 2 years after surgery. Hence, it is necessary to determine the risk factors for HCC recurrence and the markers for continuous monitoring of anti-tumor response before and after surgery. Circulating tumor cells (CTCs) is an integral part of "liquid biopsy" and has great potential to change the current treatment modality in the cancer field. CTCs are derived from solid tumors and are associated with hematogenous metastasis. Therefore, analyzing the level of CTC has clinical guiding significance. For liver cancer patients, overall survival (OS) tended to be poorer in patients with CTCs. Although surgical treatment of liver cancer has benefited most patients with liver cancer, monitoring postoperative recurrence, further improving the long-term prognosis of liver cancer, postoperative detection of CTCs and other related indicators, combined with targeted, immune and other related treatments for further study. It is expected to receive 100 patients (50 treatment groups, 50 control groups). Patients who underwent immunotherapy after surgery were assigned to the immunotherapy group, and patients who were not treated with sorafenib after surgery were classified as the control group. All patients underwent 7 CTCs tests (immunomagnetic beads negative enrichment-targeted PCR) before, 7 days after surgery and 1st, 3rd, 6th, 9th, and 12th postoperatively. All patients were observed from the observation period. After the liver cancer resection, the patient was observed to have died, lost to follow-up or the end of the study.

ELIGIBILITY:
Inclusion criteria:

* Pathological diagnosis of primary hepatocellular carcinoma, BCLC stage A,B,C, liver function Chid-Pugh grade A, or liver function Child-Pugh classification changed from grade B to grade A after short-term liver treatment, PS score 0- 1 point. Received surgical treatment of primary hepatocellular carcinoma.
* Laboratory inspection inclusion criteria:

  * Neutrophils ≥ 1.5 × 109 / L;
  * Platelets ≥ 50 × 109 / L;
  * Hemoglobin ≥ 90 g / L;
  * Serum creatinine ≤ 1.5 × upper limit of normal (ULN) and creatinine clearance ≥ 50 mL/min;
  * AST, ALT ≤ 2.5 × ULN;
  * Serum bilirubin ≤ 1.25 × ULN;
  * Patients who did not receive anticoagulant therapy: INR or aPTT ≤ 1.5 × ULN. If the patient received prophylactic anticoagulant therapy, the INR ≤ 2 × ULN within 14 days before the study treatment and the aPTT was within the normal range, the patients were acceptable for enrollment.
  * High risk factors for postoperative recurrence: Large blood vessels (2-pole branches) and bile duct invasion, or visible tumor thrombus;
  * Positive resection margin: Histopathological examination of the resected liver section indicatee residual tumor cells;
  * Two weeks after operation, AFP still ≥200 ug/L;
  * Preoperative lymph node involvement.
* General inclusion criteria:

  * Age 18-75;
  * No anti-tumor treatment history before surgery;
  * Agree to provide tissue and pathological specimens;
  * ECOG 0 points;
  * For women of gestational age, no pregnancy plan and continued full contraception.

Exclusion criteria:

* Pathological diagnosis of primary hepatocellular carcinoma, BCLC stage A, with radical resection, Child-Pugh grade C, PS score of 2 points and above. Biliary cells or mixed cell carcinoma confirmed by postoperative pathology. No surgery was performed.
* Preoperative treatment of TACE or radiotherapy and chemotherapy, and targeted anti-tumor therapy.
* One month after the operation, the rest of the anti-tumor treatment was performed, or combined with two or more anti-tumor pain treatment.
* There were distant metastases before surgery.
* Have a history of active autoimmune disease or autoimmune disease;
* Inoculated with any anti-infective vaccine (such as influenza vaccine, varicella vaccine, etc.) within 4 weeks before randomization;
* Use immunosuppressive agents, or systemic, or absorbable local hormones to achieve immunosuppressive purposes (dose > 10 mg/day of prednisone or other equivalent hormones) and continue to be used within 2 weeks prior to randomization;
* Any significant clinical and laboratory abnormalities;
* Researchers believed that the patient effected safety evaluation, such as: uncontrollable active infections, uncontrolled diabetes, high blood pressure could not be reduced to the following range by monotherapy (systolic blood pressure < 140 mmHg, diastolic blood pressure < 90 mmHg), peripheral neuropathy grade II or above, congestive heart failure, myocardial infarction within 6 months, chronic kidney disease;
* Main or main branch tumor thrombus (preoperative imaging or intraoperative findings) or extrahepatic disseminated or recurrent liver cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival | 1 year

SECONDARY OUTCOMES:
Overall Survival | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- TaoBai, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Yes